CLINICAL TRIAL: NCT00207363
Title: Does Induction PEG-Intron in Combination With Rebetol Enhance the Sustained Response Rates in Patients With Chronic Hepatitis C
Brief Title: Does Induction PEG-Intron in Combination With Rebetol Enhance the Sustained Response Rates in Patients With CHC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: T.R.U.E. Research Foundation (Unknown)
Responsible Party: Principal Investigator, Stephen A Harrison, Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2002.076
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; peginterferon alfa-2b; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial induction therapy (Experimental): Receive Peg Intron 3.0mcg/kg/wk for 12 weeks followed by Peg Intron 1.5 mcg/kg/wk for 36 weeks
  Interventions: Drug: induction therapy
- Standard of Care (Active Comparator): Peg Inter 1.5mcg/kg/wk for 48 weeks
  Interventions: Drug: Ribavirin, Peg interferon alfa 2b

INTERVENTIONS:
Drug: Ribavirin, Peg interferon alfa 2b — Peg interferon alfa 2b 1.5mcg/kg/wk for 48 weeks ribavirin 13+/-2 mg/kg daily for 48 weeks
  Other Names: Peg interferon alfa 2b (Peg Intron)
  Arms: Standard of Care
Drug: induction therapy — Peg Intron 3.0mcg/kg/wk for 12 weeks then Peg interon 1.5mcg/kg/week for 36 weeks
  Other Names: Peg Intron (peginterferon alfa 2b
  Arms: Initial induction therapy

SUMMARY:
The purpose of this study is to see which of two doses of PEG (polyethylene glycol) interferon alfa-2b in combination with Ribavirin for 48 weeks is more effective at elimination of hepatitis C.

The primary objective of this study is to compare the efficacy of Induction PEG-Interferon alfa-2b (PEG-Intron) and Ribavirin (Rebetol) to standard PEG-Interferon alfa-2b (PEG-Intron) and Ribavirin (Rebetol) in patients with chronic hepatitis C.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the use of induction dose PEG-Intron in combination with Rebetol will enhance the elimination of Hepatitis C in treatment naïve patients with genotype 1 and 4.

Currently PEG-Interferon alfa-2b plus Ribavirin results in a sustained response in 54-61% of patients with Hepatitis C. Those with genotype 1and 4 and high viral loads are the most likely to have a less favorable response. The administration of induction dose interferon in combination with Ribavirin may yield an improved sustained response rate in these more difficult to treat patients with chronic Hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* willing to give written informed consent and be able to adhere to dose and visit schedules.
* 18years of age or older of either gender and any race. Subjects who are over 65 years of age must be in generally good health.
* Serum positive for HCV-RNA by PCR assay Treatment naïve Genotype 1 & 4 HCV participants
* ALT either elevated or persistently normal
* Liver biopsy within 36 months with a pathology report confirming the histological diagnosis is consistent with CHC
* Compensated liver disease with the following minimum hematologic, biochemical, and serologic criteria at the Entry Visit

  * Hemoglobin values of <12 gm/dL for females & <13 gm/dL for males.
  * WBC <3,000/mm3
  * Neutrophil count < 1,500/mm3
  * Platelets <65,000/mm3
  * Direct bilirubin, within 20% of (ULN)
  * Indirect bilirubin, WNL (unless non-hepatitis related factors such as Gilbert's disease explain an indirect bilirubin rise
* Albumin, WNL
* Serum creatinine, within 20% of ULN
* Glucose should be less than 115 mg/dL
* Thyroid Stimulating Hormone (TSH), WNL
* HIV negative
* HBsAg negative
* Alpha fetoprotein value < 100 ng/mL obtained within one year prior to entry for patients with Stage 3 or 4 liver disease
* Reconfirmation & documentation sexually active female subjects of childbearing potential are practicing adequate contraception during the treatment period & 6 months following the last dose of study medication
* Reconfirmation that sexually active male subjects are practicing acceptable methods of contraception during the treatment period & for 6 months following the last dose of study medication

Exclusion Criteria:

* Women who are pregnant or nursing.
* Hepatitis C of non-genotype 1 or 4
* Previous anti-viral therapy
* Suspected hypersensitivity to interferon, PEG-interferon, ribavirin
* Any other cause for the liver disease other than chronic hepatitis C including but not limited to:

  * Co-infection with HBV
  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Obesity-induced liver disease
  * Drug-related liver disease
* Hemophilia or any other condition that would prevent the subject from having a liver biopsy, including anticoagulant therapy
* Hemoglobinopathies
* Evidence of advanced liver disease (ascites, bleeding varices,spontaneous encephalopathy)
* organ transplants other than cornea and hair transplant.
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of the protocol such as:Preexisting psychiatric condition, especially severe depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicidal attempt are excluded
* CNS trauma or active seizure disorders requiring medication
* Significant cardiovascular dysfunction within the past 12 months. Subjects with ECG showing clinically significant abnormalities
* Poorly controlled DM
* Chronic pulmonary disease (COPD)with documented pulmonary hypertension
* Immunologically mediated disease (e.g., inflammatory bowel disease, RA, idiopathic thrombocytopenia purpura, lupus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, clinical cryoglobulinemia with vasculitis)
* Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids
* Active gout
* Substance abuse
* not willing to be abstain from the consumption of alcohol.
* clinically significant retinal abnormalities
* Any other condition that in the opinion of the Investigator would make the subject unsuitable for enrollment, or could interfere with the subject participating in and completing the protocol
* Known HIV Positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2002-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare the efficacy of Induction PEG-Interferon alfa-2b (PEG-Intron) and Ribavirin (Rebetol) to standard PEG-Interferon alfa-2b (PEG-Intron) and Ribavirin (Rebetol) in patients with chronic hepatitis C. | 72 weeks
  Serum HCV-RNA will be evaluated at Weeks 0, 12, 24, and 48 during treatment and at Week 24 following the end of therapy. The primary efficacy endpoint is the loss of HCV-RNA at 6 months of follow up.

SECONDARY OUTCOMES:
The loss of HCV-RNA at 6 months of follow up. If the HCV-RNA has not decreased by one log at treatment week 24, the patient will be classified as a treatment nonresponder and medications are discontinued. | 72 weeks
  Serum HCV-RNA will be evaluated at Weeks 0, 12, 24, and 48 during treatment and at Week 24 following the end of therapy. The primary efficacy endpoint is the loss of HCV-RNA at 6 months of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Harrison, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Brady DE, Torres DM, An JW, Ward JA, Lawitz E, Harrison SA. Induction pegylated interferon alfa-2b in combination with ribavirin in patients with genotypes 1 and 4 chronic hepatitis C: a prospective, randomized, multicenter, open-label study. Clin Gastroenterol Hepatol. 2010 Jan;8(1):66-71.e1. doi: 10.1016/j.cgh.2009.08.036. Epub 2009 Sep 10. PMID 19747986